CLINICAL TRIAL: NCT03477825
Title: Pilot Study on the Effects of Oral Triphala and Rubia Cordifolia on the Gut Microbiome and Skin Biophysical Properties
Brief Title: Pilot Study of Triphala and Rubia Cordifolia on Gut Microbiome and Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 1174110
Record Dates: First submitted 2018-03-13; First posted 2018-03-26 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Sebum Production; Stool Microbiome; Transepidermal Water Loss; Facial Brrightness; Erythema; Wrinkles; Facial Shine
MeSH Terms: conditions — Erythema | interventions — triphala

STUDY DESIGN:
Intervention Model Description: Thirty (30) subjects meeting the inclusion criteria without any of the exclusion criteria will be enrolled in this study. This study will be a double blinded study. Each subject will be randomized a priori to receive either placebo, Rubia cordifolia, or Triphala tablets.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Group A: Placebo group (n = 10)
  * Supplement appearing similar to Herbal formulations
  * Each placebo tablet will contain microcrystalline cellulose, dicalcium phosphate, PVPK30, sodium starch glycolate, magnesium stearate, OpaDry orange coating.
  * Dose: subjects in this group will take 4 placebo tablets per day
  Interventions: Dietary Supplement: Placebo Oral Tablet
- Rubia Cordifolia (Experimental): Group B: R. cordifolia group (n = 10)
  * 2,000 mg R. cordifolia per day - supplied by Banyan Botanicals and following standard supplementation doses on commercially available supplement (https://www.banyanbotanicals.com/manjistha-tablets/)
  * Each tablet contains 500 mg of R. cordifolia per tablet.
  Interventions: Dietary Supplement: Rubia Cordifolia
- Triphala (Experimental): Group C: Triphala group (n= 10)
  * Tablets of Triphala will be supplied from Banyan Botanicals (https://www.banyanbotanicals.com/triphala-tablets-11/)
  * Each tablet contains mix Emblica officinalis, Terminalia bellerica, and Terminalia chebula
  * Dose: subjects will take 4 tablets per day, with a total dose of 2,000 mg of total herb.
  Interventions: Dietary Supplement: Triphala

INTERVENTIONS:
Dietary Supplement: Placebo Oral Tablet — Group A: Placebo group (n = 10)
  * Supplement appearing similar to Herbal formulations
  * Each placebo tablet will contain microcrystalline cellulose, dicalcium phosphate, PVPK30, sodium starch glycolate, magnesium stearate, OpaDry orange coating.
  * Dose: subjects in this group will take 4 placebo tablets per day
  Arms: Placebo
Dietary Supplement: Rubia Cordifolia — Group B: R. cordifolia group (n = 10)
  * 2,000 mg R. cordifolia per day - supplied by Banyan Botanicals and following standard supplementation doses on commercially available supplement (https://www.banyanbotanicals.com/manjistha-tablets/)
  * Each tablet contains 500 mg of R. cordifolia per tablet.
  Other Names: Manjistha
  Arms: Rubia Cordifolia
Dietary Supplement: Triphala — Group C: Triphala group (n= 10)
  * Tablets of Triphala will be supplied from Banyan Botanicals (https://www.banyanbotanicals.com/triphala-tablets-11/)
  * Each tablet contains mix Emblica officinalis, Terminalia bellerica, and Terminalia chebula
  * Dose: subjects will take 4 tablets per day, with a total dose of 2,000 mg of total herb.
  Arms: Triphala

SUMMARY:
Few studies have assessed the effects of Triphala and Rubia Cordifolia from a skin biophysical perspective. Here, we aim to understand how these herbs can modulate the skin's barrier properties and the gut microbiome.

DETAILED DESCRIPTION:
Herbal supplements such as Rubia cordifolia and Triphala [a mix of Emblica officinalis (Amalaki), Terminalia bellerica (Bibhitaki), and Terminalia chebula (Haritaki)] are commonly used for skin based treatments in India. However, the scientific evidence for their specific effects on the skin are scant. Rubia cordifolia is a root that is used in skin care for pigmentation and inflammation.1 Triphala is thought to have antioxidant properties and reduce inflammation in general. Herbs have been shown to modulate the gut microbiome, as previous studies have suggested that triphala may modify the gut microbiome.2

However, few studies have assessed the effects of these herbs from a skin biophysical perspective. Here, we aim to understand how these herbs can modulate the skin's barrier properties and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria for subjects:

1. Age 18 to 60 years of age
2. Subject must be able to read and comprehend study procedures and consent forms.

Exclusion Criteria for subjects:

1. Subject should be generally healthy and have no smoking history in the past one year.
2. Subjects must have no history of diabetes, metabolic syndrome, known cardiovascular disease, malignancy, kidney disease, or chronic steroid use.
3. Those who are unable to discontinue topical medications for two weeks.
4. Those who are unable to discontinue systemic antibiotics or oral probiotics for one month prior starting the study.
5. Those who are unable to discontinue their Triphala and Rubia Cordifolia regimen for one month prior to starting study.
6. Subjects who are postmenopausal
7. Those who are pregnant or breastfeeding
8. Those that are prisoners or cognitively impaired
9. Those who have a known allergy to Rubia cordifolia, Emblica officinalis, Terminalia bellerica, Terminalia chebula.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Sebum excretion rate | 4 weeks +/- 1 week
  Sebum production measured by sebumeter
Stool microbiome diversity via stool sample | 4 weeks +/- 1 week
  Stool microbiome diversity via stool sample

SECONDARY OUTCOMES:
Transepidermal water loss via Tewameter | 4 weeks +/- 1 week
  Transepidermal water loss via Tewameter
Facial brightness measured via photographic assessment | 4 weeks +/- 1 week
  Facial brightness measured via photographic assessment
Facial redness via photographic assessment | 4 weeks +/- 1 week
  Facial redness via photographic assessment
Facial wrinkles via photographic assessment | 4 weeks +/- 1 week
  Facial wrinkles via photographic assessment
Facial shine via photographic assessment | 4 weeks +/- 1 week
  Facial shine via photographic assessment
Digestion Questionnaire | 4 weeks +/- 1 week
  We will assess digestive symptoms such as stooling patterns and regularity based on level of frequency (Never, Sometimes, Always, Unsure).
Symptoms Questionnaire | 4 weeks +/- 1 week
  We will assess general health related symptoms based on level of frequency (Never, Sometimes, Often, Unsure).
Food Intake Log | 4 weeks +/- 1 week
  We ask for a food diary that will account for all food and drink intake in a given day for three days prior to their next visit. The diary will note what food/beverage and how much of that item was consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD, Principal Investigator — UC Davis
Locations (1):
- University of California-Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual patient data.

REFERENCES:
- [Derived] Peterson CT, Pourang A, Dhaliwal S, Kohn JN, Uchitel S, Singh H, Mills PJ, Peterson SN, Sivamani RK. Modulatory Effects of Triphala and Manjistha Dietary Supplementation on Human Gut Microbiota: A Double-Blind, Randomized, Placebo-Controlled Pilot Study. J Altern Complement Med. 2020 Nov;26(11):1015-1024. doi: 10.1089/acm.2020.0148. Epub 2020 Sep 18. PMID 32955913